CLINICAL TRIAL: NCT06238856
Title: Safety and Tolerability Study of Single Dose Escalations of TR02 (SLIT™ Amikacin) by Inhalation in Cystic Fibrosis Study Patients With Chronic Infections of Pseudomonas Aeruginosa
Brief Title: Single Dose Escalation Study of TR02 (Sustained Lipid Inhalation Technology [SLIT™] Amikacin) in Participants With Cystic Fibrosis (CF) Having Chronic Infections of Pseudomonas Aeruginosa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TR02-101
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Amikacin Dose 1 + Placebo (Experimental): Participants will receive a single dose of SLIT™ amikacin at Dose 1 or matching placebo by inhalation on Day 0.
  Interventions: Drug: SLIT™ Amikacin; Drug: Placebo
- Cohort 2: Amikacin Dose 2 + Placebo (Experimental): Participants will receive a single dose of SLIT™ amikacin at Dose 2 or matching placebo by inhalation on Day 0 upon initiation of Cohort 2.
  Interventions: Drug: SLIT™ Amikacin; Drug: Placebo
- Cohort 3: Amikacin Dose 3 + Placebo (Experimental): Participants will receive a single dose of SLIT™ amikacin at Dose 3 or matching placebo by inhalation on Day 0 upon initiation of Cohort 3.
  Interventions: Drug: SLIT™ Amikacin; Drug: Placebo

INTERVENTIONS:
Drug: SLIT™ Amikacin — Amikacin administered via the Pari LC STAR™ nebulizer.
  Other Names: TR02
Drug: Placebo — Nebulized saline.

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of three active doses of nebulized amikacin in a SLIT™ formulation.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must produce sputum that is positive for Pseudomonas aeruginosa.
* Confirmed diagnosis of CF (positive sweat chloride >60 milliequivalents (mEq)/liter (by pilocarpine iontophoresis) and/or a genotype with two identifiable mutations consistent with CF accompanied by one or more clinical features with the CF phenotype.
* Forced expiratory volume (FEV1) ≥40% predicted at Screening as calculated by the Knudsen reference equations.
* Clinically stable with no evidence of current pulmonary exacerbation.

Exclusion Criteria:

* History of lung transplantation.
* Use of intravenous antibiotics or oral quinolones within 14 days of Screening.
* Use of low dose oral antibiotics (e.g. tetracycline, sulfa) for acne or other conditions within 30 days of Screening.
* Use of systemic corticosteroids (≥20 milligrams [mg] of prednisone per day) within 30 days of Screening.
* Initiation of TOBI® (tobramycin), high dose ibuprofen, recombinant human DNase (rhDNase), or macrolide antibiotics within 60 days of Screening.
* History of sputum or throat swab culture yielding Burkholderia cepacia complex within 2 years of Screening or growth of Burkholderia cepacia complex from the sputum or throat swab culture obtained at Screening.
* History of biliary cirrhosis, portal hypertension, or splenomegaly or splenomegaly on physical exam at Screening or enrollment.
* History of daily continuous oxygen supplementation or requirement for more than 2 liter per minute (L/min) at night.

Note: Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-05-12 (Actual); Primary Completion 2005-02-08 (Actual); Study Completion 2005-02-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Experience a Treatment Emergent Adverse Event (TEAE) | Up to Day 28
  Safety and tolerability of three active doses of nebulized amikacin in a SLIT™ formulation.

SECONDARY OUTCOMES:
Area Under the Concentration-time Curve (AUC) of SLIT™ Amikacin in Serum | Pre-dose and at multiple time points post-dose up to Day 3
Percent Dose of SLIT™ Amikacin in Urine | At multiple time points post-dose up to Day 3
AUC of SLIT™ Amikacin in Sputum | Pre-dose and at multiple time points post-dose on Days 1, 2, 3, 8, 14, and 28
Change From Baseline in Sputum Density of Pseudomonas Aeruginosa | Baseline up to Day 28

IPD SHARING:
Plan to Share IPD: No